CLINICAL TRIAL: NCT06272396
Title: Feasibility and Diagnostic Relevance of Recording an ECG Trace With a Connected Watch
Brief Title: Relevance of Recording an ECG Trace With a Connected Watch
Acronym: ECG-MC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2023/64
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Arrhythmias, Cardiac
Keywords: Electrocardiogram; Smart watch; Arrhythmia; Artificial Intelligent; Remote monitoring
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smart watch (Experimental): ECG done with smart watch
  Interventions: Device: Smart watch

INTERVENTIONS:
Device: Smart watch — ECG 1D/6D

SUMMARY:
Over the past few years, various systems have been developed to record ECG traces on an ambulatory basis. The latest connected watch models feature 2-electrode ECG recording. This single (1D) or six derivations (6D) can be used to derive a wealth of information about the heart's rhythm. The information that can be derived from an ECG recording with a derivation goes far beyond̀ simple differentiation between atrial fibrillation and sinus rhythm. In contrast, in various clinical situations, a tracing restricted to an intracardiac defibrillator (ICD) may prove falsely normal, wrongly reassuring a patient and delaying management. The primary objective of the study is to evaluate the sensitivity of ECG-1D or 6D recordings from a connected watch in measuring electrical parameters, compared with a standard ECG-12D, also to obtain a bank of tracings, to create and validate an artificial intelligence algorithm for the automatic analysis of ECG tracings recorded with a connected watch and also to validate the feasibility and sensitivity of recording an ECG tracing with a connected watch in children.

DETAILED DESCRIPTION:
Single-arm prospective study to evaluate the measurement of electrocardiographic parameters obtained using two non-invasive ECG methods, one 12-lead reference method and the second 1 or 6 leads recorded from a connected watch, in a group of patients with healthy hearts (normal ECG) and 19 pathological groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized or seen in consultation in one of the departments of the Haut Lévêque cardiology hospital,
* Patient of both sexes, minor (from birth to 18 years) or adult,
* Free, informed and written consent from the patient or, in the case of minors, from the legal parent (at the latest on the day of inclusion and before any examination required for the research),
* Subject affiliated to or benefiting from a social security regime.

Exclusion Criteria:

* Person incapable of giving consent,
* Person subject to a legal protection measure (safeguard of justice, tutorship or curatorship),
* A person deprived of liberty by judicial or administrative decision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
Comparison of electrical parameters measured using the 2 ECG methods: P-wave amplitude | 36 months
  Mean of P-wave amplitude
Comparison of electrical parameters measured using the 2 ECG methods: P-wave duration | 36 months
  Mean of P-wave duration
Comparison of electrical parameters measured using the 2 ECG methods: QRS amplitude | 36 months
  Mean of QRS amplitude
Comparison of electrical parameters measured using the 2 ECG methods: QRS duration | 36 months
  Mean of QRS duration
Comparison of electrical parameters measured using the 2 ECG methods: QT/QTc | 36 months
  Mean of QT/QTc (corrected QT) intervals

SECONDARY OUTCOMES:
Creation of bank of anormal ECG trace | 36 months
  Number of ECG-1D/6D and 12 derivations
Compare the diagnostic capabilities of an ECG trace recorded with a watch against the reference method, the 12-lead ECG | 36 months
  Accuracy of diagnostic
Validate the feasibility of recording and sending of ECG tracings with a connected watch at the patient's home | 36 months
  Number of ECG-1D/6D and 12 derivations
Validate the feasibility of recording an ECG trace with a connected watch for a child | 36 months
  Number of ECG-1D/6D and 12 derivations
Validate the sensibility of an ECG trace with a connected watch for a child | 36 months
  Quality of ECG-1D/6D

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BORDACHAR, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Haut-Lévèque, Pessac, France

IPD SHARING:
Plan to Share IPD: No